CLINICAL TRIAL: NCT04681937
Title: Clinical and Radiological Comparison of the Efficacy of Hyaluronic Acid, PRP and Steroid Injections in Partial Rotator Cuff Tears: A Prospective Randomized Study
Brief Title: Comparison of Hyaluronic Acid, PRP and Steroid Injections in Partial Rotator Cuff Tears: A Prospective Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muzaffer Ağır, MD, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4350611
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Partial Tear of Rotator Cuff; Rotator Cuff Tears
Keywords: partial rotator cuff tear; subacromial injection; plateled-rich-plasma; physical therapy
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Hyaluronic Acid; Physical Therapy Modalities; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hyaluronic Acid + Physical Therapy (Experimental): 4 ml hyaluronic acid (subacromial)
  Interventions: Combination Product: Subacromial Injection (hyaluronic acid) + Physical Therapy.
- Platelet-Rich-Plasma (PRP) + Physical Therapy (Experimental): 4 ml platelet-rich-plasma (subacromial)
  Interventions: Combination Product: Subacromial Injection (Platelet-Rich-Plasma) + Physical Therapy.
- Steroid + Physical Therapy (Experimental): methylprednisolone acetate (1ml methylprednisolone acetate + 3 ml serum saline) (subacromial)
  Interventions: Combination Product: Subacromial Injection (methylprednisolone acetate) + Physical Therapy.
- Placebo (serum saline) + Physical Therapy (Experimental): 4 ml serum saline (subacromial)
  Interventions: Combination Product: Subacromial Injection (Serum Saline) + Physical Therapy.

INTERVENTIONS:
Combination Product: Subacromial Injection (hyaluronic acid) + Physical Therapy. — arm1: sodium hyaluronate (4ml) arm2: platelet-rich-plasma (4ml) arm3: methylprednisolone acetate (1ml methylprednisolone acetate + 3 ml serum saline) arm4: serum saline (4ml) The same physical therapy procedure will be applied to all arms after injection.
  Arms: Hyaluronic Acid + Physical Therapy
Combination Product: Subacromial Injection (Platelet-Rich-Plasma) + Physical Therapy. — arm1: sodium hyaluronate (4ml) arm2: platelet-rich-plasma (4ml) arm3: methylprednisolone acetate (1ml methylprednisolone acetate + 3 ml serum saline) arm4: serum saline (4ml) The same physical therapy procedure will be applied to all arms after injection.
  Arms: Platelet-Rich-Plasma (PRP) + Physical Therapy
Combination Product: Subacromial Injection (methylprednisolone acetate) + Physical Therapy. — arm1: sodium hyaluronate (4ml) arm2: platelet-rich-plasma (4ml) arm3: methylprednisolone acetate (1ml methylprednisolone acetate + 3 ml serum saline) arm4: serum saline (4ml) The same physical therapy procedure will be applied to all arms after injection.
  Arms: Steroid + Physical Therapy
Combination Product: Subacromial Injection (Serum Saline) + Physical Therapy. — arm1: sodium hyaluronate (4ml) arm2: platelet-rich-plasma (4ml) arm3: methylprednisolone acetate (1ml methylprednisolone acetate + 3 ml serum saline) arm4: serum saline (4ml) The same physical therapy procedure will be applied to all arms after injection.
  Arms: Placebo (serum saline) + Physical Therapy

SUMMARY:
There are many conservative treatment options available for partial rotator cuff tears. However, the superiority of a certain type of injection could not be demonstrated with the available data. Our aim is to compare the effectiveness of steroid, hyaluronic acid, prp and placebo (normal saline) injections in partial rotator cuff tears by applying the same physical therapy protocol after injection.

ELIGIBILITY:
Inclusion Criteria:

* persistent continous pain at least 3 months
* partial thickness rotator cuff tear on MRI

Exclusion Criteria:

* inflammatory disease
* pregnancy
* known malignancy
* bleeding disorder ( or <10 g/dl Hb level, <150.000 ul platelet)
* previous shoulder injection
* history of shoulder surgery
* full-thickness tear
* other shoulder problem (osteoarthritis, bony lesions, etc)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 12 months after injection
  minimum score:0, maximum score:100, 100 is better function.

SECONDARY OUTCOMES:
Constant-Murley Shoulder Outcome Score (CMS) | 12 months after injection
  minimum score:0, maximum score:100, 100 is better function.
Visual analogue scale (VAS) | 12 months after injection
  minimum score:0, maximum score:10, 0 is better function
Subjective Shoulder Value (SSV) | 12 months after injection
  minimum score:0, maximum score:100, 100 is better function.
Range of Motion (ROM) | 12 months after injection
  Active Shoulder Range of Motion Measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)